CLINICAL TRIAL: NCT03514043
Title: Patient and Staff Experience of Ambulatory Emergency Care on the Surgical Admissions Unit (SAU)
Status: Completed | Type: Observational
Sponsor: University of Exeter (Other)
Collaborators: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 1718/01
Record Dates: First submitted 2018-04-13; First posted 2018-05-02 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Emergencies; Surgery
Keywords: Ambulatory care; Emergency general surgery; Patient satisfaction
MeSH Terms: conditions — Emergencies; Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ambulatory care surgical patients: Patients who have attended the surgical assessment unit with an emergency general surgical condition and have their care completed without an inpatient stay.
- Surgical assessment unit staff: Staff who are involved in the care of patients on the surgical assessment unit. This includes senior and junior doctors, nurses, healthcare assistants and ward receptionists.

SUMMARY:
Emergency ambulatory care ("day-case" care that does not involve staying in a hospital bed overnight) is now well-established for medical patients and is being used increasingly for surgical patients. However, it is not known how emergency surgical patients feel about being managed in this way compared to being admitted to a hospital ward. The investigating team believe that some people will find it easier and would prefer to be able to stay at home overnight but others may find this difficult or dislike this method of care.

The investigators want to explore staff and patients' experience of this type of care with semi-structured telephone interviews. The interviews will take around 20-30mins each. The anticipated number of patient participants needed is 20 and 12-15 staff members.

DETAILED DESCRIPTION:
This is a qualitative study of patient and staff experience. Data will be collected by semi-structured telephone and face-to-face interviews.

Abdominal pain is a common reason for people to attend hospital as an emergency. It makes up a considerable proportion of the patients being admitted under the care of general surgeons. Other common reasons for people attending include infections such as abscesses and problems following previous surgery.

A Surgical Assessment Unit (SAU) is an ambulatory area with a waiting room and assessment cubicles. It is staffed by a triage nurse or healthcare assistant and doctors from the surgical team. Patients can be assessed and have investigations including blood tests and radiology procedures including x-rays, ultrasound and CT. After assessment they are either admitted to the ward, discharged home or have their care continued in an ambulatory manner returning in the next few days for further or repeat assessment.

Previously patients were either discharged or admitted for observation, investigation and treatment such as intravenous antibiotics. Many of these patients could be managed safely in a "day case" manner. This pathway allows for re-attendance should it be required.

Emergency ambulatory care is well-established in medicine for conditions such as suspected deep vein thrombosis (DVT) and transient ischaemic attack (TIA) but has not yet been widely adopted in surgery. There is uncertainty surrounding the best way of looking after these patients as the diagnosis is often uncertain and it can be difficult to judge which patients require admission.

Pilot studies have shown that up to 30% of emergency general surgical patients could be managed in this way. These studies also report a high patient satisfaction score but do not inform us what works, why and for whom. These would be important considerations for organisations looking to expand their emergency general surgical ambulatory service.

This study aims to expand upon previous work in this area by conducting semi-structured interviews with patients who have experienced emergency general surgical ambulatory care. The investigating team aim to achieve a representative sample of participants by age, attending condition and satisfaction score. They will identify themes that influence patient experience of emergency ambulatory care and whether this might vary depending on patient factors such as age, social support/responsibilities and attending condition.

Patient participants will be recruited to the study by the clinical team by means of short verbal explanation and the provision of an information sheet. Potential participants will give their contact details to be passed to the study team or will make contact themselves at a later stage. They will then by contacted by the study team and given further information over the telephone. Those wishing to proceed will have arrangements made for a telephone interview. A recording of consent will be made prior to the start of the interview and will be stored as a separate audio file.

The interview schedule has been drawn up based on areas that have emerged from work in the past using patient diaries. (Improving the Patient Experience of Ambulatory Care in the Surgical Assessment Unit, 2014) The PPI work done has included review of these questions for acceptability and ease of understanding and minor changes have been made to the wording of questions as a result. The prompts used are mainly to encourage explanations of why participants have answered the way they have.

The interviews will last 20-40mins and will be recorded using digital recording software. They will be conducted by the principal investigator. No potentially identifiable information will be recorded and participants will be advised not to divulge identifiable information prior to the interview. If this occurs inadvertently it will be deleted prior to transcription. These audio recordings will be given an anonymous identification number and then be transcribed into text documents using a paid transcription service within the UK. Once the transcription has been completed the recording will be deleted.

The transcribed data will be stored on a NHS server. It will be available for access to the study team by password protection and on request in an anonymised form by the university sponsor. Once the study is complete it will be stored on a university repository for the period required for archive and deleted from the NHS server.

The transcribed data will be coded and then undergo thematic analysis using NVIVO software. Coding will be done by the principal investigator and a proportion of the data will be separately coded by the 2 senior members of the study team. Interim analysis will be conducted after each 5 patients and the interview schedule may undergo some change to explore in more detail areas of interest that emerge.

If groups are underrepresented in the interim analysis then there may be targeted recruitment to the underrepresented group. This may include the characteristics of patient age and overall satisfaction with care given.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adult patients of any gender over the age of 18 undergoing emergency ambulatory care via the surgical assessment unit for a general surgical condition will be included.

Exclusion Criteria:

* Children under the age of 18
* Adults without capacity to consent as participants for the study

Patient participant exclusion criteria:

* Those who have primarily presented with a condition that is not within the remit of general surgeons
* Those who had their care continued as an inpatient immediately following their initial presentation.
* Unable to understand or speak English to the level required to understand the information sheet or conduct the interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults presenting to the surgical assessment unit under the care of general surgeons who have their care managed in an ambulatory manner without inpatient admission.
  Staff who are involved in the care of these patients in the groups described in the group section.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Factors affecting patient satisfaction: semi-structured interviews | Will be measured within 3 weeks of attendance
  Factors that influence patients' experience of emergency general surgical care [semi-structured interviews with patients]
Factors affecting implementation of ambulatory emergency care | Interviews will be conducted at a single timepoint from May 2019 to October 2019.
  Factors which affect how staff use ambulatory emergency care and what they perceive this issues to be with this method of care.
  This will be measured using semi-structured interviews with staff.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa H Massey, MBBS (BSc), Principal Investigator — Royal Devon and Exeter Hospital NHS Trust
Locations (1):
- Royal Devon and Exeter Hospital NHS Foundation Trust, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
At the end of the study the research data will be uploaded to an open access repository held on a University of Exeter server. Depending on practicality this may include individual participant data at interview level or may include the data post-analysis.

DOCUMENTS (1):
  • Study Protocol (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/43/NCT03514043/Prot_002.pdf